CLINICAL TRIAL: NCT05217719
Title: Effects of Recombinant Human Thrombopoietin on Platelet Levels in ICU Patients With Pneumonia With Thrombocytopenia: a Multicenter, Single-blind, Randomized Controlled Study
Brief Title: Effects of Recombinant Human Thrombopoietin on Platelet Levels in ICU Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: The Third Affiliated Hospital of Southern Medical University (Other Government); The Second People's Hospital of GuangDong Province (Other); Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Principal Investigator, Zhenhua Zen, Associate Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: nfyicu005
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Pneumonia; Thrombocytopenia
MeSH Terms: conditions — Pneumonia; Thrombocytopenia | interventions — Thrombopoietin; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the TPO group (Experimental): Patients in TPO group will be treated with rhTPO at a dose of 15000u/d, subcutaneous injection, for 7 consecutive days.
  Interventions: Drug: recombinant human thrombopoietin
- the control group (Placebo Comparator): Patients in the control group will receive the same amount of saline as a placebo, which is injected subcutaneously, for 7 consecutive days.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: recombinant human thrombopoietin — The dose of rhTPO is 15,000 U per day. The subcutaneous injection will be terminated when PCs are increased to normal. The duration of rhTPO will be 7 days.
  Arms: the TPO group
Drug: normal saline — Patients in the control group will receive the same amount of saline as a placebo, which is injected subcutaneously. The duration of saline will be 7 days.
  Arms: the control group

SUMMARY:
The incidence of thrombocytopenia in ICU patients with severe illness ranged from 8.3% to 67.6%, and ranged from 14% to 44% during ICU treatment.Severe patients with thrombocytopenia also have significantly increased bleeding events and blood transfusions, and even a significantly increased risk of death.This study examines whether elevated platelets benefit patients with pneumonia

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pneumonia (community acquired pneumonia, hospital acquired pneumonia or ventilator associated pneumonia);
* Voluntarily signed informed consent;
* ≥18 years old;
* Platelet count ≤75×109/L

Exclusion Criteria:

* A history of hematopoietic stem cell transplantation or solid organ transplantation such as liver, kidney or lung;
* Hematological malignancy;
* Immune thrombocytopenia, such as SLE, ITP, TTP, etc.
* The length of stay in ICU is less than 24h;
* Pregnant or lactation patients;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
The time to recovery to a normal platelet level | 14 days
  The clinical recovery time of platelets was defined as the time it takes to reach clinical recovery.